CLINICAL TRIAL: NCT05360030
Title: Mechanism of Analgesic Effect on Prolonged Continuous Theta Burst Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: RI2022089
Record Dates: First submitted 2022-04-19; First posted 2022-05-04 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-04

CONDITIONS: Chronic Pain; rTMS
MeSH Terms: conditions — Chronic Pain | interventions — Naloxone; Sodium Chloride; Ketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active stimulation of M1 (Experimental): pcTBS was administered to the left M1 at 80% resting motor threshold (RMT), consisting of a burst of 3 pulses given at 50 Hz repeated every 5 Hz. A total of 1,200 pulses were delivered with the TMS coil positioned in a posterior-anterior (PA) direction parallel to the midline.
  Interventions: Drug: Naloxone; Drug: Saline; Drug: Ketamine Hydrochloride; Device: pcTBS of M1
- active stimulation of DLPFC (Experimental): pcTBS was administered to the left DLPFC at 80% resting motor threshold (RMT), consisting of a burst of 3 pulses given at 50 Hz repeated every 5 Hz. A total of 1,200 pulses were delivered with the TMS coil positioned in a posterior-anterior (PA) direction parallel to the midline.
  Interventions: Drug: Naloxone; Drug: Saline; Drug: Ketamine Hydrochloride; Device: pcTBS of DLPFC
- SHAM stimulation (Sham Comparator): The Sham stimulation was delivered using the same protocol, with the coil being orientated at 90° to the scalp so that the magnetic field would be delivered away from the scal
  Interventions: Drug: Naloxone; Drug: Saline; Drug: Ketamine Hydrochloride; Device: SHAM stimulation

INTERVENTIONS:
Drug: Naloxone — The volunteer received an intravenous bolus followed by a continuous infusion of naloxone, which was continued throughout the pcTBS session
Drug: Saline — The volunteer received an intravenous bolus followed by a continuous infusion of placebo (saline), which was continued throughout the pcTBS session
Drug: Ketamine Hydrochloride — The volunteer received an intravenous bolus followed by a continuous infusion of ketamine, which was continued throughout the pcTBS session
Device: pcTBS of M1 — Prolonged continuous theta-burst stimulation (pcTBS) was administered to the left M1 at 80% RMT, consisting of a burst of 3 pulses given at 50 Hz repeated every 5 Hz. A total of 1,200 pulses were delivered with the TMS coil positioned in a posterior-anterior (PA) direction parallel to the midline
  Arms: active stimulation of M1
Device: pcTBS of DLPFC — Prolonged continuous theta-burst stimulation (pcTBS) was administered to the left DLPFC at 80% RMT, consisting of a burst of 3 pulses given at 50 Hz repeated every 5 Hz. A total of 1,200 pulses were delivered with the TMS coil positioned in a posterior-anterior (PA) direction parallel to the midline
  Arms: active stimulation of DLPFC
Device: SHAM stimulation — The Sham stimulation was delivered using the same pcTBS protocol, with the coil being flipped 90◦to the scalp so that the magnetic field would be delivered away from the scalp
  Arms: SHAM stimulation

SUMMARY:
It has been shown that prolonged continuous theta burst stimulation (pcTBS) , a relatively new repetitive transcranial magnetic simulation (rTMS) protocol, of the primary motor cortex (M1) or dorsolateral prefrontal cortex (DLPFC) decreases pain in healthy volunteers, in various experimental models. In addition, rTMS of M1 has also been shown to have analgesic effects in various chronic pain conditions, including neuropathic pain.The mechanisms underlying rTMS-induced analgesia remain unclear. Functional neuroimaging studies have shown that rTMS of M1 and DLPFC induces changes in the activity of cortical and subcortical structures involved in pain processing and modulation. Endogenous opioids and e N-methyl-D-aspartate (NMDA) receptor are known to play a major role in these processes. The investigator hypothesized that the endogenous opioids systems (EOS) and NMDA receptor might be involved in the analgesic action of pcTBS. In the first part,the investigator compares the analgesic effects of motor cortex (M1) or dorsolateral prefrontal cortex (DLPFC) stimulation before and after naloxone or placebo treatment, the intensity of pain induced by capsaicin were used to evaluate the analgesic effects of pcTBS. If naloxone does not reverse the analgesic effect of pcTBS,The volunteers will be invited to participant the second part of the study, which the investigator compares the analgesic effects of motor cortex (M1) or dorsolateral prefrontal cortex (DLPFC) stimulation before and after Ketamine treatment.

DETAILED DESCRIPTION:
This study comprised 3 parallel arms corresponding to 3 types of stimulation: active stimulation of M1, active stimulation of DLPFC-pcTBS, and sham stimulation (of M1 or DLPFC). Volunteers were randomly assigned to the 3 arms. In the first part, these volunteers participated in 2 experimental sessions 1 weeks apart, in which we compared the effects of naloxone and placebo (saline), administered according to a randomized, double-blind crossover design, on pcTBS-induced analgesia. Each experimental session started with the determination of baseline pain intensity and cortical excitability as well as plasma opioid peptide concentrations. Ten minutes before pcTBS (of M1, DLPFC, or sham), the volunteer received an intravenous bolus followed by a continuous infusion of either placebo (ie, saline) or naloxone, which was continued throughout the rTMS session (2 minutes). The participant was then allowed to rest for 60 minutes. Posttreatment pain intensity, cortical excitability and plasma opioid peptide concentrations will be determined by the same procedure used at baseline.In the second part, ketamine will be delivered the same as the first part.

ELIGIBILITY:
Inclusion Criteria:

1）woman or man over 18 and under 85 years old; 2）Clinical diagnosis of physical and mental health people; 3) able to cooperate in completing questionnaire.

Exclusion Criteria:

1)Clinical diagnosis of psychiatric disorder including major depression; 2) History of substance abuse (alcohol, drugs); 3) Past treatment with repetitive transcranial magnetic stimulation (rTMS); 4) Contraindications to rTMS (previous severe head trauma or neurosurgical intervention, past or current epilepsy, active brain tumor, intracranial hypertension, implanted ferromagnetic devices, e.g., cardiac pacemaker, neurostimulator, or cochlear implants); 5) Any difficulty to fill out questionnaires (due to language or cognitive problems);

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-05-14 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
pain intensity at baseline | Baseline
  pain intensity on a 10-cm visual analogue scale (VAS) extending from 0 (no pain) to 100 (maximal pain possible) at baseline.
pain intensity at the posttreatment of pcTBS | through study completion, an average of 8 months
  pain intensity on a 10-cm visual analogue scale (VAS) extending from 0 (no pain) to 100 (maximal pain possible) at the posttreatment of pcTBS.

SECONDARY OUTCOMES:
Motor-evoked potential (MEP) | through study completion, an average of 8 months
  Corticospinal excitability will be measured with MEP at rest of the first dorsal interosseous (FDI) muscle, A total of 20 single pulses were consecutively delivered to the hand region of the left M1 at 120% RMT (45° to the midline, handle pointing backward).
Cortical silent period (CSP) | through study completion, an average of 8 months
  Corticospinal excitability will be measured with CSP during a sustained voluntary FDI muscle contraction, A total of 20 single pulses were consecutively delivered to the hand region of the left M1 at 120% RMT (45° to the midline, handle pointing backward).
Maximum plasma concentration of opioid peptide at baseline | baseline
  plasma opioid peptide concentrations will be measured using ELISA at baseline.
Maximum plasma concentration of opioid peptide at the posttreatment of pcTBS | through study completion, an average of 8 months
  plasma opioid peptide concentrations will be measured using ELISA at the last posttreatment of pcTBS.

CONTACTS AND LOCATIONS:
Overall Officials: min yan, prof, Study Chair — The second affiliated hospital of Zhejiang University hangzhou
Locations (1):
- The second affiliated hospital of Zhejiang University hangzhou, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Sun J, Wu C, Ren J, He Y, Sun N, Huang H, Chen Q, Liu D, Huang Y, Xu F, Yu L, Fitzgibbon BM, Cash RFH, Fitzgerald PB, Yan M, Che X. Characterizing the opioidergic mechanisms of repetitive transcranial magnetic stimulation-induced analgesia: a randomized controlled trial. Pain. 2024 Sep 1;165(9):2035-2043. doi: 10.1097/j.pain.0000000000003220. Epub 2024 Mar 26. PMID 38537053